CLINICAL TRIAL: NCT05050695
Title: Relationship Between Lumbopelvic Muscles Activity and Ultrasonographic Measurement of Contralateral Anterior Humeral Translation in Chronic Unilateral Low Back Pain
Brief Title: Correlation Between Posterior Oblique Sling Activation and Contralateral Glenohumeral Stability in Low Back Pain
Status: Completed | Type: Observational
Sponsor: Shaimaa Ramadan Ibrahim Abdul-ghani El Deab (Other)
Responsible Party: Sponsor-Investigator, Shaimaa Ramadan Ibrahim Abdul-ghani El Deab, Assistant lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/001843
Record Dates: First submitted 2021-09-11; First posted 2021-09-20 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with unilateral chronic low back pain: Subjects with low back pain for more than 3 months on one side of the spine
- Healthy subjects: Subjects without a history of low back pain

SUMMARY:
Objective: This study will be conducted to investigate the relationship between the amplitude of posterior oblique sling muscles; ipsilateral gluteus maximus (GM) and contralateral latissmus Dorsi (LD), and the amount of anterior translation of humeral head (ATHH) of the contralateral glenohumeral joint (GHJ) in subjects with unilateral chronic low back pain (CLBP) during ipsilateral prone knee extension (PHE) test. Methods: The study will be conducted on thirty subjects (15 patients with CLBP and 15 healthy subjects). Ipsilateral GM and contralateral LD amplitude will be recorded by surface EMG during PHE of the limb at the painful side and correlated to ATHH of contralateral GHJ as measured by ultrasonography. Hypothesis: There won't be a significant relationship between the amplitude of posterior oblique sling muscles (GM and contralateral LD) during PHE for the ipsilateral leg and the amount of ATHH of the contralateral GHJ in patients with unilateral CLBP.

DETAILED DESCRIPTION:
Demographic data will be collected from all subjects regarding age, weight, height, and body mass index. After patient selection according to the inclusion and exclusion criteria, measuring the amplitude of gluteus maximus (GM) and contralateral latissmus dorsi (LD) muscles during prone hip extension (PHE) for the ipsilateral leg to the symptoms in unilateral CLBP patients and for the selected leg in matched controls will be carried out using surface electromyography (EMG) unit. Then ultrasonography unit will be used to assess the amount of anterior translation of humeral head (ATHH) of contralateral glenohumeral joint for both groups.

Before placement of the EMG electrodes, the skin at the anatomic landmarks will be shaved (if required), rubbed, and cleaned with isopropyl alcohol 70% to remove excess oils and debris.

The electrodes will be sterilized and placed on the muscle belly oriented parallel to the muscle fiber away from the tendon and muscle edges with the inter-electrodes distance of two centimeters. The electrodes will be secured by adhesive tape. Before recording, skin impedance will be checked to be less than 5 KΩ.

The electrodes for LD will be placed 4 cm below the inferior tip of the scapula and half the distance between the spine and the lateral edge of the torso. For GM, electrodes will be placed at half the distance between the greater trochanter and second sacral vertebra and at an oblique angle at, or slightly above, the level of the trochanter.

The two normalization procedures will be the typical maximal voluntary isometric contraction (MVIC) performed as per SENIAM Guidelines (www.seniam.org), and submaximal voluntary contraction (sub-MVC) task will be performed using the prone double leg raise. It is recommended to avoid maximal contractions of the GM muscle, because reproduction of pain on testing would have possibly invalidated the use of the root mean square (RMS) values for normalization.

For the sub-MVC of GM, the subjects will be asked to lift both knees 5 cm off the examination table while the knees should be flexed at 90 and held them for 5 seconds in a prone position. Three trials will be performed with 30 seconds rest in between.

For MVIC of LD muscle, the subjects will be in prone position and the side being tested is aligned with the edge of the plinth, with the shoulder and upper extremity off the plinth. The subjects will be asked to flex the elbow and manual isometric resistance will be applied at distal humerus during shoulder extension and adduction and the contraction held for 5 seconds, the middle 3 seconds will be used for the analysis. Stabilization will be applied to the ipsilateral scapula and trunk. Three trials were performed with 30 seconds rest in between.

For recording during PHE, all subjects will be instructed about active PHE and The target angle was set at 10 degrees to control the amount of hip extension using a goniometer. A 30 seconds rest period will be provided between each trial.

Ultrasonography assessment: the patient will be assessed in a sitting position and the shoulder will be placed in internal rotation then the position will be maintained by a sling. Two therapists are needed to assess humeral translation.

ELIGIBILITY:
Inclusion Criteria for CLBP group:

1. Patients age between 20-50yrs
2. Patients with chronic low back pain (pain > 3 months).
3. Patients with unilateral symptoms (facet, disc, SIJ dysfunction) will be referred by an orthopedic physician with or without referral to the leg.

Inclusion Criteria for the healthy control group:

1. matched controls in terms of age, weight, height, and BMI.

Exclusion Criteria for both groups:

1. History of shoulder pain 3 months ago.
2. History of any shoulder pathology.
3. Congenital pathology affecting the spine or shoulder.
4. Any neurological disorder.
5. Non-mechanical LBP (e.g., fracture, malignancy, infection)
6. Difficulty performing the PHE task because of weakness in the GM or the test provokes pain.
7. BMI 30 or higher as fat tissue may decrease the ability to measure surface EMG activity

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients with CLBP will be recruited from the orthopedic outpatient clinic at Kasr El Ainy hospital and the outpatient clinic of the faculty of physical therapy, Cairo University.
  Healthy subjects will be recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Amplitude of gluteus maximus muscle | From admission to discharge, up to two weeks
  Investigator will collect the EMG activity of gluteus maximus during PHE using two silver surface recording electrodes for bipolar configuration
Amplitude of latissimus dorsi muscle | From admission to discharge, up to two weeks
  Investigator will collect the EMG activity of latissimus dorsi during PHE using two silver surface recording electrodes for bipolar configuration
Anterior translation of humeral head | From admission to discharge, up to two weeks
  Investigators will assess the anterior humeral translation using ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Bassem G. El Nahass, Professor, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No